CLINICAL TRIAL: NCT01385423
Title: Haploidentical Donor Natural Killer (NK) Cell Infusion With Intravenous Recombinant Human IL-15 (rhIL-15) in Adults With Refractory or Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: Haploidentical Donor Natural Killer Cell Infusion With IL-15 in Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010LS063; MT2010-10 (Other: Blood and Bone Marrow Transplantation Program); 1009M89012 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: acute myelogenous leukemia; natural killer cells; haploidentical donor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine phosphate; Cyclophosphamide; Interleukin-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- IL-15 Patients with AML (Experimental): Adults with Refractory or Relapsed Acute Myelogenous Leukemia (AML) treated with preparative regimen and Intravenous Recombinant Human IL-15 (rhIL-15)
  Interventions: Drug: Preparative Regimen; Biological: Intravenous Recombinant Human IL-15 (rhIL-15)

INTERVENTIONS:
Drug: Preparative Regimen — Fludarabine 25 mg/m^2 x 5 days start day -6, Cyclophosphamide 60 mg/kg x 2 days on day -5 and -4 (*if < 4 months from prior transplant, omit day -4 dose)
  Other Names: Fludara; Cytoxan
Biological: Intravenous Recombinant Human IL-15 (rhIL-15) — IL-15 at assigned dose (0.25, 0.5, 0.75 1, 2 and 3 mcg/kg for 3 to 6 patients) intravenously (IV) over 30 minutes once a day beginning day +1 and continuing for 12 doses
  Other Names: IL-15

SUMMARY:
This is a single center, "modified standard design" dose escalation study designed to determine the maximum tolerated, minimum efficacious dose (MTD/MED) of IL-15 (Intravenous Recombinant Human IL-15) and incidence of donor natural killer (NK) cell expansion by day +14 when given after haploidentical donor NK cells in patients with relapse or refractory acute myelogenous leukemia (AML).

DETAILED DESCRIPTION:
Once the MTD/MED for IL-15 is determined, this cohort will be expanded to a total of 19 patients. The primary goal of this extended phase will be to establish a correlation of the clinical endpoint, CRp defined as leukemic clearance (< 5% marrow blast and no peripheral blood blasts) and neutrophil recovery without platelet recovery, with in vivo expansion.

Patients achieving a complete remission and neutrophil recovery (ANC > 500) for at least 4 weeks will be considered for allogeneic transplant to prolong remission independent of this study.

All patients, including those who go on to transplant, will be followed to determine disease free survival, treatment related mortality, and time to relapse.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Meets one of the following disease criteria:

  * Primary acute myelogenous leukemia (AML) induction failure: no complete response (CR )after 2 or more induction attempts
  * Relapsed AML or Secondary AML (from MDS or treatment-related): not in CR after 1 or more cycles of standard induction therapy. For patients > 60 years of age the 1 cycle of standard chemotherapy is not required if either of the following is met:
* relapse within 6 months of last chemotherapy
* blast count <30% within 10 days of starting protocol

  * AML relapsed > 2 months after transplant who do not have the option of donor lymphocyte infusions (e.g. recipients of autologous or umbilical cord blood [UCB] transplants)

Patients with prior central nervous system (CNS) involvement are eligible provided that it has been treated and cerebrospinal fluid (CSF) is clear for at least 2 weeks prior to enrollment. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.

* Available related HLA-haploidentical donor (3-5 of 6 HLA-A, B and C)
* Karnofsky Performance Status > 50%
* Adequate organ function defined as:

  * Creatinine: ≤ 2.0 mg/dL
  * Hepatic: Liver function tests (LFT's) < 5 times upper limit of institutional normal (ULN)
  * Pulmonary Function: oxygen saturation ≥ 90% on room air and pulmonary function >50% corrected DLCO and FEV1 Testing required only if symptomatic or prior known impairment.
  * Cardiac Function: Ejection fraction (EF) ≥ 40%, no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to Natural Killer (NK) cell infusion (excluding preparative regimen pre-medications)
* Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy.
* Voluntary written consent

Exclusion Criteria:

* Bi-phenotypic acute leukemia
* Transplant < 60 days prior to study enrollment
* Pregnant or breastfeeding - The agents used in this study include those that fall under Pregnancy Category D - have known teratogenic potential. Women of child bearing potential must have a negative pregnancy test within 14 days of study treatment start
* Active autoimmune disease
* History of severe asthma, presently on chronic medications (a history of mild asthma not requiring therapy is eligible)
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that has not been evaluated with bronchoscopy, if feasible. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections). Surgical resection waives any waiting requirements.
* Uncontrolled bacterial or viral infections - chronic asymptomatic viral hepatitis is allowed
* Pleural effusion large enough to be detectable on chest x-ray
* Known hypersensitivity to any of the study agents used
* Received investigational drugs within the 14 days before enrollment
* Known active CNS involvement

Criteria For Initial Donor Selection:

* Related donors (sibling, parent, offspring, parent or offspring of an HLA identical sibling)
* 14-75 years of age
* At least 40 kilogram body weight
* In general good health as determined by the evaluating medical provider
* HLA-haploidentical donor/recipient match (low resolution)
* Not pregnant
* Agree to undergo donor viral screening panel
* Able and willing to undergo apheresis
* Voluntary written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated/Minimum Efficacious Dose | Day 42
  Determine the maximum tolerated, minimum efficacious dose (MTD/MED) of recombinant human IL-15; dose limiting toxicity (DLT) occurring during the first 42 days after the NK cell infusion; MED = if 2 of 3 patients or 4 of 6 patients has an in vivo NK cell count >2500, then dose escalation with cease as it will be in the range of a biologic dose which may achieve the goal of in vivo expansion without pushing IL-15 doses higher to toxicity.

SECONDARY OUTCOMES:
Incidence of Expansion of Natural Killer Cells | Day 14 after Infusion
  defined by measuring an absolute circulating donor-derived NK cell count of >100 cells/μl in the patient's peripheral blood by day +14 after the NK cell infusion.
Treatment Related Mortality (TRM) | Day 1 of Treatment until Day of Death
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Rate of CRp | Day 28-42
  defined as leukemia clearance (< 5% marrow blasts and no peripheral blood blasts) and neutrophil recovery without platelet recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cooley S, He F, Bachanova V, Vercellotti GM, DeFor TE, Curtsinger JM, Robertson P, Grzywacz B, Conlon KC, Waldmann TA, McKenna DH, Blazar BR, Weisdorf DJ, Miller JS. First-in-human trial of rhIL-15 and haploidentical natural killer cell therapy for advanced acute myeloid leukemia. Blood Adv. 2019 Jul 9;3(13):1970-1980. doi: 10.1182/bloodadvances.2018028332. PMID 31266741